CLINICAL TRIAL: NCT04209244
Title: Effect of Fish Oil Versus Placebo on Hyperlipidemia and Toxicities in Children and Young Adults With Acute Lymphoblastic Leukemia - A Randomized Controlled Trial
Brief Title: Effect of Fish Oil on Hyperlipidemia and Toxicities in Children and Young Adults With Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Child Cancer Foundation (Other)
Responsible Party: Principal Investigator, Renate Dagsdottir Laumann, Principal Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-19054660
Record Dates: First submitted 2019-12-19; First posted 2019-12-24 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Leukemia, Acute Lymphoblastic
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Fish Oils; Rapeseed Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fish oil (Experimental): Eskimo-3 Pure Fish Oil, 10 ml per day (2.6 g EPA+DHA)
  Interventions: Dietary Supplement: Eskimo-3 Pure Fish Oil
- Placebo (Placebo Comparator): Rapeseed Oil, 10 ml per day
  Interventions: Dietary Supplement: Rapeseed Oil

INTERVENTIONS:
Dietary Supplement: Eskimo-3 Pure Fish Oil — Dosage: 10 ml/day (2.6 g EPA+DHA)
  Other Names: Fish Oil
  Arms: Fish oil
Dietary Supplement: Rapeseed Oil — Dosage: 10 ml/day (0 g EPA+DHA)
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Acute lymphoblastic leukemia (ALL) is the most common malignant disease among children. Treatment results have improved over time due to intensive risk-adapted therapy and the 5-year survival rate is now above 90%. However, the burden of therapy has increased proportionally. Many children develop serious acute and chronic side effects, which impact on the patients expected lifespan and impair their quality of life as a result of therapy. Treatment with PEG-asparaginase and dexamethasone increases the levels of triglycerides and total cholesterol. Consequently, the incidence of hyperlipidemia is high during initial ALL therapy. Studies have suggested that hyperlipidemia is a risk factor for development of osteonecrosis, thrombosis and possibly acute pancreatitis.

Long-chained marine omega-3 fatty acids, found in fish oil, decrease levels of triglycerides and total cholesterol in hyperlipidemic patients. Due to the high survival rate, it is of great interest to develop methods to reduce treatment related toxicities.

The investigators hypothesise that daily intake of fish oil will prevent development of hyperlipidemia during ALL treatment phases with dexamethasone and PEG-asparaginase compared to placebo and that fish oil intake may reduce the incidence of severe adverse events related to ALL treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children (1-17.9 years) and young adults (18-45 years) diagnosed with ALL, stratified to very-low risk (VRL), intermediate risk low (IR-low) and intermediate risk high (IR-high) in the ALLTogether protocol.

Exclusion Criteria:

* Patients diagnosed with ALL, stratified to high risk (HR) after induction treatment or stem cell transplantation in the ALLTogether protocol

Ages: 1 Year to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-12-16 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Hyperlipidemia | From treatment day 4 until treatment day 169 or 204
  Triglycerides and/or total cholesterol levels five times or more than the age-dependent upper normal limit.

SECONDARY OUTCOMES:
Lipid metabolism | VLR and IR-low: 4, 11, 18, 25, 32, 39, 46, 53, 60, 67, 81, 95, 109, 123, 137, 151 and 169. IR-high: treatment day 4, 11, 18, 25, 32, 39, 46, 53, 60, 67, 74, 81, 88, 95, 102, 109, 123, 137, 151, 165, 179, 193 and 204.
  Triglycerides, total cholesterol, VLDL-cholesterol, LDL-cholesterol and HDL-cholesterol.
Compliance | From treatment day 4 until end of intervention (treatment day 169 or 204)
  Assessed by self-registration forms, return of bottles and levels of EPA+DHA in whole blood
Bone density | DEXA-scan at start and end of intervention. Bone biomarkers at treatment day 4, 81 and 169 for VLR and treatment day 4, 102 and 204 for IR-low and IR-high.
  Assessed by DEXA-scan and bone biomarkers (iCa, PTH, vit D, phosphate, magnesium, creatinine, alkaline phosphatase, CTX, P1NP.
Hemostatic status | At treatment day 4, 81 and 169 for VLR and at treatment day 4, 102 and 204 for IR-low and IR-high
  Thromboelastography (TEG), multiplate and thrombocytes.
Endothelial function | At treatment day 4, 81 and 169 for VLR and at treatment day 4, 102 and 204 for IR-low and IR-high
  sTM, syndecan-1, PECAM, VEGFR1
Incidence of severe adverse events | From treatment day 4 until end of intervention (treatment day 169 or 204)
  Cumulative incidence of osteonecrosis, asparaginase associated pancreatitis and thrombosis.

OTHER OUTCOMES:
Milder side effects | At end of intervention (day 169 or 204)
  Assessed by questionnaire.
Dietary intake | At treatment day 4, 81 and 169 for VLR and at treatment day 4, 102 and 204 for IR-low and IR-high
  Assessed by 3-day food records

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Leth Frandsen, Study Chair — Rigshospitalet, Denmark
Locations (4):
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No